CLINICAL TRIAL: NCT01476774
Title: NORSPAN Transdermal Patches Phase III Study In Non-Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma (China) Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BP08-CN-001
Record Dates: First submitted 2011-11-17; First posted 2011-11-22 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Disease (or Disorder); Intervertebral Disc, With Myelopathy (Manifestation)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buprenorphine Transdermal System (Active Comparator)
  Interventions: Drug: Buprenorphine Transdermal System
- Tramadol CR (Active Comparator)
  Interventions: Drug: Buprenorphine Transdermal System

INTERVENTIONS:
Drug: Buprenorphine Transdermal System — Titration period（21 days）:BTDS 5 mg or oral tramadol CR 100 mg bid, and will then be titrated, if necessary, a maximum of BTDS 20 mg or oral tramadol CR 200 mg bid will be given.
  maintenance period(5 week):Patients will continue at a dosage level that provided acceptable pain control .
  Arms: Tramadol CR
Drug: Buprenorphine Transdermal System — Titration period（21 days）:BTDS 5 mg or oral tramadol CR 100 mg bid, and will then be titrated, if necessary, a maximum of BTDS 20 mg or oral tramadol CR 200 mg bid will be given.
  maintenance period(5 week):Patients will continue at a dosage level that provided acceptable pain control .
  Arms: Buprenorphine Transdermal System

SUMMARY:
This is a multiple-dose, double-blind, double-dummy, active-control, parallel-group, multi-center, safety and efficacy study.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age are ≥20 ,≤80 years.
* Clinical diagnosis of musculoskeletal pain for 4 weeks or longer with non-malignant pain etiology at Visit 1.
* Subject is a current user of NSAIDS or paracetamol and reports a history of insufficient therapeutic benefit in musculoskeletal pain.
* Subjects must record an 'average pain over the last week at study institution' score at primary pain site of ≥ 4 on an 11-point numerical pain rating scale.
* Subjects must be able to understands the study procedures and assessment, and agree to participate in the study by giving written informed consent.

Exclusion Criteria:

* Subjects who have been taking long-acting or short-acting opioid analgesic formulations within the last 4 weeks.
* Subjects who have a current chronic disease(s) or who have a past history and high possibilities to relapse, in addition to their musculoskeletal pain, requiring frequent analgesic therapy.
* Subjects with clinically unstable respiratory disease, dysfunction of the biliary tract, thyroid disease, adrenal cortical insufficiency, prostatic hypertrophy requiring intervention or renal artery stenosis.
* Subject who have a past history of malignant neoplasm including leukemia and lymphoma.
* Subjects with clinically unstable, active or symptomatic heart disease.
* Subjects who have psychiatric disorder, uncontrolled seizures or convulsive disorder and so on.
* Subjects who have a current or past (within 5 years) history of substance or alcohol abuse, or subjects who give a positive result in drug abuse test during the Screening Period.
* Subjects scheduled for therapies within the study period which might effect study assessment.
* Females who are pregnant, lactating or have a possibility of being pregnant.
* Subjects with values > 2 times the upper limit of normal for AST or ALT or total bilirubin at visit 1 or who have severe impaired liver function.
* Subjects with serum creatinine > 2 mg/dL at Visit 1 or who have severe impaired renal function.
* Subjects with serum potassium < 3.5 mEq/L at Visit 1.
* Subjects receiving hypnotics or other central nervous system (CNS) depressants.
* Subjects receiving monoamine oxidase inhibitor (MAOI) within 2 weeks before screening.
* Subjects who have a history of supersensitivity to study drug.
* Known intolerance to and/or lack of effect of tramadol.
* Subjects who participated in a clinical research study within 1 month of study entry.
* Subjects who participated previously in a BTDS study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary Efficacy Variable is the change of Pain Intensity (Patients Visual Analogue Scale) from baseline | 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mundipharma China Ltd., Study Chair — Mundipharma China Ltd.
Locations (1):
- Investigational Site:Peking Union Medical Hospital (PUMC), Beijing, China

REFERENCES:
- [Derived] Leng X, Li Z, Lv H, Zheng Y, Liu Y, Dai K, Yao C, Yan X, Zeng X. Effectiveness and Safety of Transdermal Buprenorphine Versus Sustained-release Tramadol in Patients With Moderate to Severe Musculoskeletal Pain: An 8-Week, Randomized, Double-Blind, Double-Dummy, Multicenter, Active-controlled, Noninferiority Study. Clin J Pain. 2015 Jul;31(7):612-20. doi: 10.1097/AJP.0000000000000144. PMID 25503600